CLINICAL TRIAL: NCT03111654
Title: A Pilot Study on the Prevention of the Vascular RISK Related to Atrial Fibrillation After Intracranial Hemorrhage by Closing the Left Auricle
Acronym: RIVAFAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PI2016_843_0005
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Intracranial Hemorrhages
MeSH Terms: conditions — Atrial Fibrillation; Intracranial Hemorrhages

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with pericardial closure of the auricle (Other)
  Interventions: Diagnostic Test: Compare the risk of a vascular event
- Patients without closure of the auricle (Other)
  Interventions: Diagnostic Test: Compare the risk of a vascular event

INTERVENTIONS:
Diagnostic Test: Compare the risk of a vascular event — Collected in a post-stroke follow-up consultation, patient clinical outcome data, functional and cognitive disability, standardized, using validated scales.
  Analysis of selected therapeutic options for the prevention of AF ischemic events.

SUMMARY:
Atrial fibrillation (AF) is a frequent heart rhythm disorder, responsible for the formation of cardiac thrombi, which can embolize in the systemic circulation, responsible for strokes (Cerebrovascular accidents). AF increases the risk of stroke and stroke-related disability. Preventing the thromboembolic risk associated with FMD is therefore a public health issue. The reference treatment is oral anticoagulation but this treatment is contraindicated in patients with a history of intracranial hemorrhage. The percutaneous closure of the auricle is a recent technique which makes it possible to exclude this appendix from the left atrium where the majority of thrombi are formed in the framework of the AF. Comparative studies have shown the effectiveness of this technique, appearing to be similar to that of anticoagulation. However, in view of the per-procedural risk, the indication of closure was retained by the health authorities only in the event of a contraindication to oral anticoagulants in patients with non-valvular AF with a high thromboembolic risk. Patients with a history of intracranial hemorrhage are therefore candidates for this technique, but there are few studies where these patients were included. The risk-benefit must be demonstrated over the long term, in terms of ischemic, hemorrhagic recurrence and becoming functional and cognitive.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Affiliation to a social security scheme
* Non-valvular, paroxysmal, persistent or permanent atrial fibrillation
* CHA2DS2-VASc greater than or equal to 2
* History of intracranial haemorrhage: Intra-parenchymal hematoma, subacute or chronic subcutaneous hematoma And
* Patients having benefited from the percutaneous closure of the auricle at the University Hospital of Amiens
* Either patient admitted to the CHU of Amiens in neurology, neurosurgery or geriatrics for intracranial haemorrhage, who received standard medical treatment for the comparison group.

Exclusion Criteria:

* CHADS2VASC2 less than 2
* Extradural hematoma
* Arachnoidal haemorrhage by rupture of aneurysm
* Haemorrhagic transformation of ischemic stroke
* Other indication of anticoagulation than FA
* Modified Rankin scale greater than 4 following intracranial hemorrhage.
* Early death, in the month following the onset of intracranial hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Compare the risk of vascular event (ischemic stroke, haemorrhagic stroke, systemic embolism or cardiovascular or indeterminate death) in patients treated at the Amiens University Hospital with a history of AF and intracranial haemorrhage | 1 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France